CLINICAL TRIAL: NCT04937387
Title: A Phase III, 12 Week, Randomized, Double-blind, 4 Arm Parallel Group Bridging Study, Comparing the Efficacy, Safety and Tolerability of the Fixed Dose Combination FF/UMEC/VI Once-daily Via a Dry Powder Inhaler With Dual Combination of FF/VI, Administered in Chinese Participants With Inadequately Controlled Asthma
Brief Title: Efficacy and Safety of Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI) in Chinese Participants With Inadequately Controlled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 214263
Record Dates: First submitted 2021-06-02; First posted 2021-06-24 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Asthma; Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI); Fluticasone Furoate/Vilanterol (FF/VI); ELLIPTA; Chinese
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Participants receiving FF/VI at Dose level 1 via ELLIPTA inhaler (Experimental)
  Interventions: Drug: FF/VI; Device: ELLIPTA
- Cohort 2: Participants receiving FF/UMEC/VI at Dose level 2 via ELLIPTA inhaler (Experimental)
  Interventions: Drug: FF/UMEC/VI; Device: ELLIPTA
- Cohort 3: Participants receiving FF/ VI at Dose level 3 via ELLIPTA inhaler (Experimental)
  Interventions: Drug: FF/VI; Device: ELLIPTA
- Cohort 4: Participants receiving FF/UMEC/VI at Dose level 4 via ELLIPTA inhaler (Experimental)
  Interventions: Drug: FF/UMEC/VI; Device: ELLIPTA

INTERVENTIONS:
Drug: FF/VI — FF/VI will be administered.
  Arms: Cohort 1: Participants receiving FF/VI at Dose level 1 via ELLIPTA inhaler; Cohort 3: Participants receiving FF/ VI at Dose level 3 via ELLIPTA inhaler
Drug: FF/UMEC/VI — FF/UMEC/VI will be administered.
  Arms: Cohort 2: Participants receiving FF/UMEC/VI at Dose level 2 via ELLIPTA inhaler; Cohort 4: Participants receiving FF/UMEC/VI at Dose level 4 via ELLIPTA inhaler
Device: ELLIPTA — FF/UMEC/VI and FF/VI will be administered via ELLIPTA inhaler.

SUMMARY:
The study aims to evaluate the efficacy, safety and tolerability of FF/UMEC/VI compared with FF/VI via ELLIPTA® inhaler in Chinese participants with inadequately controlled asthma. ELLIPTA is a registered trademark of GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 years or older at the time of signing the informed consent.
* Documented history asthma diagnosis as defined by the Global Initiative for Asthma (GINA) at least one year prior to Visit 0.
* Participants with inadequately controlled asthma (ACQ-6 score >=1.5) despite Inhaled Corticosteroids/Long-Acting Beta-2-Agonists (ICS/LABA) maintenance therapy at Visit 1.
* Participants who require daily ICS/LABA for at least 12 weeks prior to Visit 0 with no changes to maintenance asthma medications during the 6 weeks immediately prior to Visit 0 (including no changes to a stable total dose of ICS of greater than [>]250 micrograms (mcg) per day fluticasone propionate [FP, or equivalent]).
* A best pre-bronchodilator morning (AM) FEV1 >=30 percent (%) and less than (<) 85% of the predicted normal value at Visit 1. Predicted values will be based upon the European Respiratory Society (ERS) Global Lung Function Initiative.
* Airway reversibility defined as >=12% and >=200 milliliters (mL) increase in FEV1 between 20 and 60 minutes following 4 inhalations of albuterol/salbutamol aerosol at Visit 1.
* All participants must be able to replace their current Short-Acting Beta-2-Agonists (SABA) inhaler with albuterol/salbutamol aerosol inhaler at Visit 1 as needed for the duration of the study. Participants must be judged capable of withholding albuterol/salbutamol for at least 6 hours prior to study visits.
* Male or female participants following contraceptive/barrier requirements and it should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of non-childbearing potential (WONCBP) or a woman of childbearing potential (WOCBP) who agrees to follow the contraceptive guidance during the study.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Chest X-ray documented pneumonia in the 6 weeks prior to Visit 1.
* Any asthma exacerbation requiring a change in maintenance asthma therapy in the 6 weeks prior to Visit 1.
* Participants with the diagnosis of chronic obstructive pulmonary disease, as per Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines, including all of the following:

  1. History of exposure to risk factors (especially tobacco smoke, occupational dusts and chemicals, smoke from home cooking and heating fuels).
  2. A post-albuterol/salbutamol FEV1/Forced Vital Capacity (FVC) ratio of <0.70 and a post-albuterol/salbutamol FEV1 of less than or equal to (<=)70% of predicted normal values.
  3. Onset of disease >=40 years of age.
* Participants with current evidence of pneumonia, active tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases or abnormalities other than asthma.
* Immune suppression (e.g., Human Immunodeficiency virus [HIV], Lupus) or other risk factors for pneumonia (e.g., neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis). Participants at potentially high risk (e.g., very low Body Mass Index [BMI], severely malnourished, or very low FEV1) will only be included at the discretion of the Investigator.
* Participants with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Unstable liver disease as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Clinically significant Electrocardiogram (ECG) abnormality: Evidence of a clinically significant abnormality in the 12-lead ECG performed during screening. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the participant's medical history and exclude participants who would be at undue risk by participating in the trial. An abnormal and clinically significant finding is defined as a 12-lead tracing that is interpreted as, but not limited to, any of the following:

  1. Atrial Fibrillation with rapid ventricular rate >120 beats per minute (bpm).
  2. Sustained or non-sustained ventricular tachycardia.
  3. Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted).
  4. QT interval corrected for heart rate by Fridericia's formula (QTcF) >=500 milliseconds (msec) in participants with QRS <120 msec and QTcF >=530 msec in participants with QRS >=120 msec.
* Participants with any of the following at Screening (Visit 1):

  1. Myocardial infarction or unstable angina in the last 6 months.
  2. Unstable or life-threatening cardiac arrhythmia requiring intervention in the last 3 months.
  3. New York Heart Association (NYHA) Class IV Heart failure [American Heart Association, 2016].
* Participants with a medical condition such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy or bladder neck obstruction should only be included if in the opinion of the Investigator the benefit outweighs the risk and that the condition would not contraindicate study participation.
* Participants with carcinoma that has not been in complete remission for at least 5 years. Participants who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the participant has been considered cured by treatment.
* Participants with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Participants who are medically unable to withhold their albuterol/salbutamol for the 6-hour period required prior to spirometry testing at each study visit.
* Participants who are:

  1. Current smokers (defined as participants who have used inhaled tobacco products within the 12 months prior to Visit 1, e.g. cigarettes, electronic-cigarettes/vaping, cigars or pipe tobacco).
  2. Former smokers with a smoking history of >=10 pack years (e.g. >=20 cigarettes per day for 10 years).
* Participants with a known or suspected history of alcohol or drug abuse within the last 2 years.
* A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate.
* Participants at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Study Investigators, sub-Investigators, study coordinators, employees of a participating Investigator or study site, or immediate family members of the aforementioned that is involved with this study.
* In the opinion of the Investigator, any participant who is unable to read and/or would not be able to complete study related materials.

Inclusion criteria for randomization:

* Participants with inadequately controlled asthma (ACQ-6 score >=1.5) at Visit 2.
* A best pre-bronchodilator morning (AM) FEV1 >=30% and <90% of the predicted normal value at Visit 2. Predicted values will be based upon the ERS Global Lung Function Initiative (Quanjer).
* Liver function tests at Visit 1:

  1. Alanine aminotransferase (ALT) <2 times upper limit of normal (ULN).
  2. Alkaline phosphatase <=1.5 times ULN.
  3. Bilirubin <=1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Compliance with completion of the Electronic diary reporting defined as completion of all questions/assessment on >=4 of the last 7 days during the run-in period.

Exclusion criteria for randomization:

* Occurrence of a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear during the run-in period that led to a change in asthma management or, in the opinion of the Investigator, is expected to affect the participant's asthma status or the participant's ability to participate in the study.
* Evidence of a severe exacerbation during screening or the run-in period, defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids.
* Changes in asthma medication (excluding run-in medication and albuterol/salbutamol inhalation aerosol provided at Visit 1).
* Evidence of clinically significant abnormal laboratory tests during screening or run-in which are still abnormal upon repeat analysis and are not believed to be due to disease(s) present. Each Investigator will use his/her own discretion in determining the clinical significance of the abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (44):
- China (44):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Dongguan
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Guilin
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Hohhot
  - GSK Investigational Site, Huizhou
  - GSK Investigational Site, Jiangmen
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Kunming
  - GSK Investigational Site, Lanzhou
  - GSK Investigational Site, Lianyungang
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Nanning
  - GSK Investigational Site, Qingdao
  - GSK Investigational Site, Qingyuan
  - GSK Investigational Site, Qinhuangdao
  - GSK Investigational Site, Sanya
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Shenzhen
  - GSK Investigational Site, Shijiazhuang
  - GSK Investigational Site, Taiyuan
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Ürümqi
  - GSK Investigational Site, Wenzhou
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Wuxi
  - GSK Investigational Site, Xi'an
  - GSK Investigational Site, Xiamen
  - GSK Investigational Site, Xinxiang
  - GSK Investigational Site, Xuzhou
  - GSK Investigational Site, Yinchuan
  - GSK Investigational Site, Zhanjiang
  - GSK Investigational Site, Zhengzhou
  - GSK Investigational Site, Zhongshan
  - GSK Investigational Site, Zunyi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 359 participants were randomized, however 1 participant was randomized in error and did not receive any study intervention. Therefore, 358 participants were included in 'Intent to Treat (ITT)' Population.
Groups:
- Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug: Participants with inadequately controlled asthma received a single dose of 100 ug fluticasone furoate [FF] and 25 ug vilanterol [VI] as a dual dose combination in a single inhaler (ELLIPTA) via inhalation for 12 weeks.
- Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug: Participants with inadequately controlled asthma received a single dose of 100 ug fluticasone furoate [FF] /62.5 ug umeclidinium [UMEC] /25 ug vilanterol [VI] as a fixed dose combination in a single inhaler (ELLIPTA) via inhalation for 12 weeks.
- Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug: Participants with inadequately controlled asthma received a single dose of 200 ug Fluticasone Furoate [FF] and 25 ug Vilanterol [VI] as a dual dose combination in a single inhaler (ELLIPTA) via inhalation for 12 weeks.
- Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug: Participants with inadequately controlled asthma received a single dose of 200 ug Fluticasone Furoate [FF]/ 62.5 ug umeclidinium [UMEC] / 25 ug Vilanterol [VI] as a fixed dose combination in a single inhaler (ELLIPTA) via inhalation for 12 weeks.
Period: Overall Study
Arm/Group | Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug
Started | 91 | 90 | 89 | 89
Safety (Safety population included all randomized participants who took at least 1 dose of study intervention.) | 90 | 90 | 89 | 88
Intent to Treat (ITT) Population (Intent to Treat (ITT) Population included all randomized participants, excluding those who were randomized in error.) | 91 | 90 | 89 | 88
Completed | 88 | 90 | 86 | 86
Not Completed | 3 | 0 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1
Not completed — Randomized in error | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population includes all randomized participants, excluding-those who were randomized in error.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug | Total
Number analyzed (Participants) | 91 | 90 | 89 | 88 | 358
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (11.5) | 52.6 (11.22) | 50.7 (12.23) | 49.9 (12.19) | 51.6 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 48 | 52 | 58 | 209
  Male | 40 | 42 | 37 | 30 | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian- East Asian Heritage | 91 | 90 | 89 | 88 | 358

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12 (100ug FF)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on treatment is defined as the highest FEV1 value obtained prior to the morning dose of investigational product. Baseline value is the latest acceptable assessment with non-missing value at the randomization visit (Visit 2).
Time Frame: Baseline (pre-dose at Day 1) and Week 12
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants who received 100ug FF, excluding those who were randomized in error and did not receive the study drug. Only those participants with data available at specified time points have been analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug
Number analyzed (Participants) | 83 | 87
Liters | 0.078 (0.0321) | 0.136 (0.0316)
Statistical Analysis 1: Comparison: Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug; Test type: Other; Least Squares Mean Difference = 0.059, 95% CI 2-sided [-0.030 to 0.147], Standard Error of Mean 0.0449; Analysis performed using mixed effect model for repeated measures with covariates of treatment, age, sex, eCRF-reported pre-study ICS dosage at screening (med, high), baseline trough FEV1 value, visit, and interaction terms for baseline trough FEV1-by-visit and treatment-by-visit, covariance structure = unstructured
Statistical Analysis 2: Comparison: Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug; Test type: Other; Posterior Mean = 0.076, 90% CI 2-sided [0.025 to 0.115] — Analysis was conducted in the Bayesian paradigm using the pre-specified mixture prior distribution, which was updated with the treatment difference between FF/UMEC/VI 100/62.5/25 and FF/VI 100/25 estimated in the MMRM analysis
Statistical Analysis 3: Comparison: Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug; Test type: Other; Posterior Median = 0.079, 95% CI 2-sided [0.005 to 0.123] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Change From Baseline in Trough FEV1 at Week 12 (200ug FF)
Description: as for outcome 1
Time Frame: Baseline (pre-dose at Day 1) and Week 12
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants who received 200ug FF, excluding those who were randomized in error and did not receive the study drug. Only those participants with data available at specified time points have been analyzed
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug
Number analyzed (Participants) | 84 | 82
Liters | 0.121 (0.0319) | 0.116 (0.0325)
Statistical Analysis 1: Comparison: Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug; Test type: Other; Least Squares Mean Difference = -0.005, 95% CI 2-sided [-0.094 to 0.084], Standard Error of Mean 0.0455; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug; Test type: Other; Posterior Mean = 0.023, 90% CI 2-sided [-0.071 to 0.103] — Analysis was conducted in the Bayesian paradigm using the pre-specified mixture prior distribution, which was updated with the treatment difference between FF/UMEC/VI 200/62.5/25 and FF/VI 200/25 estimated in the MMRM analysis
Statistical Analysis 3: Comparison: Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug; Test type: Other; Posterior Median = 0.023, 95% CI [-0.086 to 0.110] — [estimate comment as in outcome 2, analysis 2]

3. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-7) Total Score at Week 12
Description: ACQ-7 is a 7-item questionnaire to assess asthma control in participants. Six attributes are measured with a patient-completed questionnaire, and the questions are designed to be self-completed by the participant. The six patient-reported questions enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions consist of a zero (no impairment/limitation) to six (total impairment/ limitation) scale. The recall period is the past week. The seventh attribute of the ACQ-7 is lung function (FEV1%-predicted) which was assessed via study visit spirometry. All 7 items of ACQ have response on 0-6 ordinal scale (0=no impairment/limitation, 6=total impairment/limitation). The total score is calculated as the average of all non-missing item responses, ranges from 0 to 6. Higher score indicates worst symptoms.
Time Frame: Baseline (pre-dose at Day 1) and Week 12
Population: ITT population. Intent-to-Treat (ITT) Population comprised of all randomized participants, excluding those who were randomized in error and did not receive the study drug. Only those participants with data available at specified time points have been analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug
Number analyzed (Participants) | 83 | 86 | 84 | 81
Scores on a scale | -0.940 (0.0586) | -0.968 (0.0579) | -0.926 (0.0584) | -0.814 (0.0595)
Statistical Analysis 1: Comparison: Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug; Test type: Other; Least Squares Mean Difference = -0.028, 95% CI 2-sided [-0.190 to 0.134], Standard Error of Mean 0.0823; Analysis performed using mixed effect model for repeated measures with covariates of treatment, age, sex, eCRF-reported pre-study ICS dosage at screening (med, high), baseline ACQ-7 total score, visit, and interaction terms for baseline ACQ-7 total score-by-visit and treatment-by-visit, covariance structure = unstructured
Statistical Analysis 2: Comparison: Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug vs Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug; Test type: Other; Least Squares Mean Difference = 0.112, 95% CI 2-sided [-0.052 to 0.276], Standard Error of Mean 0.0832; [other analysis details as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality, Non-serious AEs and serious AEs were collected up to approximately 12 weeks.
Description: Data for All-Cause Mortality was collected for the ITT Population (all randomized participants, excluding those who were randomized in error). Serious and Other (Not Including Serious) Adverse Events were collected for the Safety Population (all randomized participants who received at least 1 dose of study intervention [any component]).
Arm/Group | Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug | Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/90 | 0/89 | 0/88
Serious Adverse Events (participants affected / at risk) | 2/90 | 3/90 | 3/89 | 1/88
Other Adverse Events (participants affected / at risk) | 16/90 | 18/90 | 22/89 | 18/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug (N=90) | Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug (N=90) | Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug (N=89) | Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug (N=88)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial bridging (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Furoate [FF] 100 Microgram[ug] / Vilanterol [VI] 25 ug (N=90) | Fluticasone Furoate [FF] 100 ug/ Umeclidinium [UMEC] 62.5 ug/ Vilanterol [VI] 25 ug (N=90) | Fluticasone Furoate [FF] 200 ug / Vilanterol [VI] 25 ug (N=89) | Fluticasone Furoate [FF] 200 ug/ Umeclidinium [UMEC] 62.5 ug/Vilanterol [VI] 25 ug (N=88)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 7 (7) | 10 (15) | 4 (4)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3) | 5 (5) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (3) | 3 (3) | 4 (5) | 4 (4)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (5) | 3 (5)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04937387/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT04937387/SAP_001.pdf